CLINICAL TRIAL: NCT01837264
Title: Phase I, Arteriocyte Magellan MAR01 Therapy - Compartment Syndrome and Battlefield Trauma Study Protocol
Brief Title: Phase I, Arteriocyte Magellan MAR01 Therapy - Compartment Syndrome and Battlefield Trauma
Acronym: Magellan MAR01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arteriocyte, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ART-11-003
Record Dates: First submitted 2013-04-17; First posted 2013-04-23 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-01

CONDITIONS: Compartment Syndrome
Keywords: Magellan MAR01; Autologous Platelet Rich Plasma; Compartment Syndrome; Battlefield Trauma; Fasciotomy
MeSH Terms: conditions — Compartment Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bone Marrow Cell Concentrate (Experimental)
  Interventions: Device: Magellan®

INTERVENTIONS:
Device: Magellan®
  Other Names: autologous cell concentrate; autologous Bone Marrow Cell Concentrate Using the Magellan® System

SUMMARY:
Compartment syndrome (CS) is a condition resulting from increased pressure within a compartment, which compromises circulation and can lead to critical limb ischemia. CS is one of the biggest medical challenges that our soldiers face after battlefield related injuries. Chronic or exercise-induced compartment syndrome (CS)rarely requires treatment; acute compartment syndrome is a medical emergency requiring surgery. Treatment of compartment syndrome is limited to fasciotomy, which relieves the pressure.The study purpose is to evaluate the feasibility and safety of the administration of marrow-derived autologous bone marrow concentrate and PRP gel generated by a point of care marrow separation system for the treatment of compartment syndrome. And to show this treatment possibly enhances wound healing, bone healing, perfusion, infection control, and the return of limb function in patients with CS.

Stem Cell and regenerative medicine development efforts for therapeutic angiogenesis and wound healing have predominantly focused on the mechanism of action of a single stem cell population to achieve neovascularization and improve tissue perfusion. It is well documented that other cells, including platelets, are efficient carriers of growth factors (VEGF-PDGF, bFGF, and SDF-1) and play active roles in angiogenesis and wound healing. Arteriocyte's development efforts focus on concentration of autologous bone marrow-derived stem cells and platelets for delivery to the site of injury in a concentration sufficient to effect local tissue revascularization and repair. These products provide for the rapid, bedside preparation of autologous PRP and bone marrow stem cell concentrate.

This clinical trial with the Magellan® System is for the preparation of autologous cell concentrate for the treatment of wound, tissue and bone healing, improved perfusion, infection control, and the return of limb function in patients at risk of amputation.

ELIGIBILITY:
Inclusion Criteria:

* Is able to provide signed, written informed consent prior to study entry
* Speaks English
* compartment fasciotomy of tibial compartment
* Sufficient skin for primary closure
* Is male or female, 18 - 65 years of age
* ABI less than 0.7, ankle pressure < 50 mmHg, or toe pressure < 30 mmHg.
* TcPO2 < 40 mmHg.
* Female subjects must be of non childbearing potential (defined as postmenopausal for at least 1 year or surgically sterile [bilateral tubal ligation, bilateral oophorectomy or hysterectomy]) or must be using adequate contraception (practicing one of the following methods of birth control):

Total abstinence from sexual intercourse (minimum of one complete menstrual cycle before study entry), A partner who is physically unable to impregnate the subject (e.g., vasectomized)Contraceptives (oral, parenteral, or transdermal) for 3 consecutive months prior to patient's cell concentrate administration, Intrauterine device (IUD), or Double barrier method (condoms, sponge, diaphragm, or vaginal ring with spermicidal jellies or cream)

* If female of childbearing potential, subject must have a negative urine pregnancy test at screening
* Confirmation of age-appropriate cancer screening consistent with the American Cancer Society guidelines.

Exclusion Criteria:

* Prior compartment syndrome fracture of same limb
* Previous fracture of the same limb
* Any contraindication to stem cell or platelet-rich plasma therapy.
* Pregnancy
* Have an active malignancy or have undergone treatment for a malignancy in the preceding 5 years, with the exception of successful treatment of non-melanoma skin cancer.
* Stage 4 or greater chronic kidney disease (eGFR < 30 ml/min, MDRD estimate).
* Unwilling or unable to comply with follow-up visits.
* Is unable to refrain from nicotine, caffeine and alcohol for a period beginning 24 hours prior to the treatment visit
* Has received an investigational medication or other study trial participation within 30 days prior to the Treatment Visit
* Prisoner
* Non-English Speaker

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-01; Primary Completion 2016-09 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Time to treatment failure or death | 12 months
  * Measurement of rate of infection in the study population
  * Complications due to wound and/or therapy
  * Amputation of limb and/or death

SECONDARY OUTCOMES:
Perfusion and quality of life measurements | 12 months
  Wound healing (rate and qualitative healing assessment)
  * Bone healing (Radiographic assessment)
  * Tissue perfusion (ABI; TcPO2)
  * Limb pain (pain score assessment)
  * Functional performance vs. uninjured limb

CONTACTS AND LOCATIONS:
Overall Officials: Brian Barnes, PhD, Study Director — Arteriocyte, Inc.
Locations (1):
- Advocate Christ Medical Center, Oak Lawn, Illinois, United States

REFERENCES:
- [Background] Ritenour AE, Dorlac WC, Fang R, Woods T, Jenkins DH, Flaherty SF, Wade CE, Holcomb JB. Complications after fasciotomy revision and delayed compartment release in combat patients. J Trauma. 2008 Feb;64(2 Suppl):S153-61; discussion S161-2. doi: 10.1097/TA.0b013e3181607750. PMID 18376159
- [Background] Ateschrang A, Ochs BG, Ludemann M, Weise K, Albrecht D. Fibula and tibia fusion with cancellous allograft vitalised with autologous bone marrow: first results for infected tibial non-union. Arch Orthop Trauma Surg. 2009 Jan;129(1):97-104. doi: 10.1007/s00402-008-0699-2. Epub 2008 Aug 2. PMID 18677497
- [Background] Sebecic B, Gabelica V, Patrlj L, Sosa T. Percutaneous autologous bone marrow grafting on the site of tibial delayed union. Croat Med J. 1999 Sep;40(3):429-32. PMID 10411974
- [Background] Umemura T, Nishioka K, Igarashi A, Kato Y, Ochi M, Chayama K, Yoshizumi M, Higashi Y. Autologous bone marrow mononuclear cell implantation induces angiogenesis and bone regeneration in a patient with compartment syndrome. Circ J. 2006 Oct;70(10):1362-4. doi: 10.1253/circj.70.1362. PMID 16998273
- [Background] Middleton S, Clasper J. Compartment syndrome of the foot--implications for military surgeons. J R Army Med Corps. 2010 Dec;156(4):241-4. doi: 10.1136/jramc-156-04-07. PMID 21275358
- [Background] Lenk K, Adams V, Lurz P, Erbs S, Linke A, Gielen S, Schmidt A, Scheinert D, Biamino G, Emmrich F, Schuler G, Hambrecht R. Therapeutical potential of blood-derived progenitor cells in patients with peripheral arterial occlusive disease and critical limb ischaemia. Eur Heart J. 2005 Sep;26(18):1903-9. doi: 10.1093/eurheartj/ehi285. Epub 2005 Apr 26. PMID 15855189
- [Background] Melillo E, Ferrari M, Balbarini A, Pedrinelli R. Transcutaneous oxygen and carbon dioxide levels with iloprost administration in diabetic critical limb ischemia. Vasc Endovascular Surg. 2006 Aug-Sep;40(4):303-11. doi: 10.1177/1538574406291824. PMID 16959724